CLINICAL TRIAL: NCT06406023
Title: Effectiveness of Instrument Assisted Soft Tissue Mobilization in Management of Piriformis Syndrome
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 01795
Record Dates: First submitted 2024-04-18; First posted 2024-05-09 (Actual); Last update posted 2024-05-09 (Actual); Status verified 2024-05

CONDITIONS: Piriformis Syndrome
MeSH Terms: conditions — Piriformis Muscle Syndrome

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Instrument assisted soft tissue mobilization (Experimental): IASTM with Graston tool along with conventional treatment in first 6 sessions. Apply hot pack for 10 mins on low back as passive warm up then AROM's of Hip (5 reps x 2 sets each) will be performed. Apply Graston tool at 30-60 degrees angle along the length of following muscles Piriformis, Gluteus medius and Hamstrings after applying emollient for 40-120 seconds.
  Piriformis stretch, SLR, Sciatic nerve stretch (3 reps x 20 sec hold x 2 sets/3 days/week for 2 weeks).
  Only Conventional protocol will be followed for remaining 6 sessions. 3 days/ week for 2 weeks. Hot pack will be applied for 10 minutes on low back followed by Strengthening exercises of Hip abductors (Hip abduction with band in sitting, standing, side-lying hip raise), and hip extensors (Gluteal bridges, Prone hip extension, Prone hams curl). (5 reps x 2 sets each/3 days/week for 2 weeks).
  Interventions: Other: Conventional treatment; Other: Instrument assisted soft tissue mobilization
- Conventional Treatment (Other): Only conventional treatment will be given in this group. Stretching exercises for 6 sessions and strengthening exercises for remaining 6 sessions.
  For first 6 sessions, hot pack will be applied for 10 minutes on low back. AROM's of Hip (5 reps x 2 sets each/ 3 days/week for 2 weeks). Piriformis stretch 3 reps x 20 sec hold x 2 sets/ 3 days/week for 2 weeks. SLR (5reps x 10 sec hold x 2 sets/ 3 days/ week for 2 weeks). Sciatic nerve stretch (5 reps x 10 sec hold x 2 sets/ 3 days/ week for 2 weeks).
  In next 6 sessions, strengthening exercises will be performed after applying hot pack on low back for 10 minutes in each session. Hip abductors strengthening (Hip abduction with band in sitting, standing, side-lying hip raise) 5reps x 2 sets each/ 3 days/ week for 2 weeks, and hip extensors (Gluteal bridges, Prone hip extension, Prone hams curl). (5 reps x 2 sets each/ 3 days/ week for 2 weeks).
  SLR (5 reps x 10 sec hold x 2 sets 3 days/ week for 2 weeks).
  Interventions: Other: Conventional treatment

INTERVENTIONS:
Other: Conventional treatment — Hot pack will be applied for 10 minutes. AROM's of Hip (5 reps x 2 sets each). Piriformis stretch 3 reps x 20 sec hold x 2 sets. SLR (5reps x 10 sec hold x 2 sets). Sciatic nerve stretch (5 reps x 10 sec hold x 2 sets) for 3 days/ week for 2 weeks.
  Strengthening exercises will be performed after 2 weeks of previous intervention of Hip abductors (Hip abduction with band in sitting, standing, side-lying hip raise), and hip extensors (Gluteal bridges, Prone hip extension, Prone hams curl). (5 reps x 2 sets each).
  SLR (5 reps x 10 sec hold x 2 sets) each exercise will be performed 3 days/ week for 2 weeks.
  Total treatment protocol will be followed for 4 weeks. Each session will be of 30 minutes.
Other: Instrument assisted soft tissue mobilization — Instrument assisted soft tissue mobilization IASTM with Graston tool along with conventional treatment in first 6 sessions. Apply hot pack for 10 mins on low back as passive warm up then AROM's of Hip (5 reps x 2 sets each) will be performed. Apply Graston tool at 30-60 degrees angle along the length of following muscles Piriformis, Gluteus medius and Hamstrings after applying emollient for 40-120 seconds.
  Arms: Instrument assisted soft tissue mobilization

SUMMARY:
This study aims to assess the effectiveness of IASTM on pain, ROM, Disability and Quality of life among Piriformis Syndrome patients. This study will add to the growing body of knowledge as there are very limited researches done in Pakistan using IASTM in patients with Piriformis Syndrome.

DETAILED DESCRIPTION:
Instrument assisted soft tissue mobilization (IASTM) is a skilled intervention that includes the use of specialized tools to manipulate the skin, myofascia, muscles, and tendons by various direct compressive stroke techniques. It has neurophysiological effect as it stimulates mechanosensitive neurons through skin deformation by using instrument. IASTM affects the vascular response to the injured soft tissue, through increasing the blood flow, reduce the stress and strain to the injured areas, decrease inflammation, increase muscle flexibility and strength, increase blood flow, break up scar tissue, promote proper tissue repair, enhance functional movements, accelerates fibroblast activity.

In 2022 there is a study that stated the overall Prevalence of piriformis muscle syndrome which is 18.3%. The Mean±SD of exact BMI were 27.43±6.859. Male and female Pace sign were 14.2% and 18.3% positive respectively.

Positive Prevalence of piriformis muscle syndrome in the general population in Age groups chi-square value is (47.753b) and P- Value (<0.001).

A 2018 study determined that Hip abductor and extensor strengthening along with neural mobilization and piriformis stretching have significant effect on improving hip abductor strength and lower extremity function when compared with neural mobilization and piriformis stretching alone in patients with Piriformis syndrome.

Another study conducted in 2022, showed the effects of IASTM in discogenic Sciatica along with neural mobilization and lumbar traction and concluded that IASTM alleviated pain and impairments in patients with sciatic nerve entrapment. Whereas, this study will assess the effectiveness of IASTM in non discogenic causes of piriformis syndrome.

A 2016 study showed the efficacy of manual therapy interventions for improving the signs and symptoms of carpal tunnel syndrome by comparing 2 manual therapy techniques: Graston Instrument-assisted soft tissue mobilization (GISTM) and soft tissue mobilization for mild to moderate cases of CTS. Results shows improvements in both groups with pain, nerve conduction latencies, wrist strength and ROM. This study will only assess the effectiveness of IASTM on pain, ROM, disability and quality of life among patients with piriformis syndrome.

Reference article showed efficacy by comparing 2 manual therapy techniques, GISTM and STM in management of carpal tunnel syndrome. There is significant improvement in wrist strength and ROM with IASTM application as it increases muscle flexibility and strength, improves blood flow, breaks up adhesions, reduce stress to injured area, enhance functional movements, increase fibroblastic activity and decreases inflammation. Current study will only assess effectiveness of IASTM on pain, ROM, functional disability and QOL among patients with piriformis syndrome. No evidence in previous studies shows efficacy of IASTM with Graston tool in management of piriformis syndrome. Hence, this study will show effectiveness of IASTM on pain, ROM, disability and quality of life in patients with piriformis syndrome.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed patients of Piriformis syndrome.
* Only females will be included in this study.
* Participants aged 30-65 years.
* Pain due to non-discogenic sciatic nerve entrapment in sub gluteal space.
* Pain aggravated by prolonged sitting, lying, standing.
* Positive FAIR test, Pace sign, Laseque sign, Beatty maneuver and Freiberg test.
* Negative Kemp sign, Milgram's test, Bowstring test, Braggard test and Lasegue differential test.

Exclusion Criteria:

* Patients with any Intrinsic Etiology such as Haemarthrosis, rheumatoid arthritis or infection.
* Patients with any recent severe trauma, fractures, subluxation or ligament injury.
* Malignancy, Open wound Fracture, DVT, Compartment syndrome, Pregnancy.
* Patients with irreversible nerve damage.
* Patients with lumbar disc herniation or any disc pathology.

Ages: 30 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Tool will be applied on Piriformis, Hamstrings and Gluteus medius muscles. Considering ethical values only female participants will be included in this study.
Enrollment: 38 (Estimated)
Dates: Start 2024-01-10 (Actual); Primary Completion 2024-06-30 (Estimated); Study Completion 2024-06-30 (Estimated)

PRIMARY OUTCOMES:
Lower Extremity Functional Scale (LEFS) | 4th week
  It is a questionnaire containing 20 questions about a person's ability to perform everyday tasks. The LEFS can be used by clinicians as a measure of patients' initial function, ongoing progress and outcome, as well as to set functional goals. The LEFS can be used to evaluate the functional impairment of a patient with a disorder of one or both lower extremities or to monitor the patient over time and to evaluate the effectiveness of an intervention. This scale scores ranges from 0-80 on a 5 point Likert scale. Changes from baseline, 2nd and 4th week LEFS will be taken.
12 item Short Form Survey (SF-12) | 4th week
  It is a self-reported outcome measure assessing the impact of health on an individual's everyday life. It is often used as a quality of life measure. The SF-12 is a shortened version of its predecessor, the SF-36. It consists of 12 item questions measuring quality of life. Changes from baseline, 2nd and 4th week SF-12 will be taken.
Sciatica Bothersomeness Index (SBI) | 4th week
  It is used to measure the participants' level of sciatica. The scale's ratings range from 0 to 6, with higher levels indicating severe sciatica discomfort. Changes from baseline, 2nd and 4th week SBI will be taken.

SECONDARY OUTCOMES:
NPRS | 4th week
  The Numerical Pain Rating Scale (NPRS) is a subjective measure in which individuals rate their pain on an eleven-point numerical scale. The scale is composed of 0 (no pain at all) to 10 (worst imaginable pain). NPRS is the most commonly used version which has good test-retest reliability. Changes from baseline, 2nd week and 4th week NPRS will be taken.
ROM of Hip Flexion | 4th week
  Changes from baseline, 2nd week and 4th week Hip flexion will be taken with goniometer.
ROM of Hip Abduction | 4th week
  Changes from baseline, 2nd week and 4th week Hip abduction will be taken with goniometer.
ROM of Hip Internal Rotation | 4th week
  Changes from baseline, 2nd week and 4th week Hip internal rotation will be taken with goniometer.

CONTACTS AND LOCATIONS:
Overall Officials: Ramsha Tariq, Masters, Principal Investigator — Senior Lecturer
Locations (1):
- Railway General Hospital, Rawalpindi, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Cass SP. Piriformis syndrome: a cause of nondiscogenic sciatica. Curr Sports Med Rep. 2015 Jan;14(1):41-4. doi: 10.1249/JSR.0000000000000110. PMID 25574881
- [Background] Kim J, Sung DJ, Lee J. Therapeutic effectiveness of instrument-assisted soft tissue mobilization for soft tissue injury: mechanisms and practical application. J Exerc Rehabil. 2017 Feb 28;13(1):12-22. doi: 10.12965/jer.1732824.412. eCollection 2017 Feb. PMID 28349028
- [Background] Seffrin CB, Cattano NM, Reed MA, Gardiner-Shires AM. Instrument-Assisted Soft Tissue Mobilization: A Systematic Review and Effect-Size Analysis. J Athl Train. 2019 Jul;54(7):808-821. doi: 10.4085/1062-6050-481-17. Epub 2019 Jul 19. PMID 31322903
- [Background] Burke J, Buchberger DJ, Carey-Loghmani MT, Dougherty PE, Greco DS, Dishman JD. A pilot study comparing two manual therapy interventions for carpal tunnel syndrome. J Manipulative Physiol Ther. 2007 Jan;30(1):50-61. doi: 10.1016/j.jmpt.2006.11.014. PMID 17224356
- [Background] Ahmad Siraj S, Dadgal R. Physiotherapy for Piriformis Syndrome Using Sciatic Nerve Mobilization and Piriformis Release. Cureus. 2022 Dec 26;14(12):e32952. doi: 10.7759/cureus.32952. eCollection 2022 Dec. PMID 36712711
- [Background] Cheatham SW, Stull KR, Kolber MJ. Roller massage: is the numeric pain rating scale a reliable measurement and can it direct individuals with no experience to a specific roller density? J Can Chiropr Assoc. 2018 Dec;62(3):161-169. PMID 30662071
- [Background] Jones A, Sealey R, Crowe M, Gordon S. Concurrent validity and reliability of the Simple Goniometer iPhone app compared with the Universal Goniometer. Physiother Theory Pract. 2014 Oct;30(7):512-6. doi: 10.3109/09593985.2014.900835. Epub 2014 Mar 25. PMID 24666408
- [Background] Grovle L, Haugen AJ, Keller A, Natvig B, Brox JI, Grotle M. The bothersomeness of sciatica: patients' self-report of paresthesia, weakness and leg pain. Eur Spine J. 2010 Feb;19(2):263-9. doi: 10.1007/s00586-009-1042-5. Epub 2009 Jun 2. PMID 19488793
- [Background] Binkley JM, Stratford PW, Lott SA, Riddle DL. The Lower Extremity Functional Scale (LEFS): scale development, measurement properties, and clinical application. North American Orthopaedic Rehabilitation Research Network. Phys Ther. 1999 Apr;79(4):371-83. PMID 10201543
- [Background] Webster KE, Feller JA. Comparison of the short form-12 (SF-12) health status questionnaire with the SF-36 in patients with knee osteoarthritis who have replacement surgery. Knee Surg Sports Traumatol Arthrosc. 2016 Aug;24(8):2620-6. doi: 10.1007/s00167-015-3904-1. Epub 2016 Jan 28. PMID 26821809